CLINICAL TRIAL: NCT01352000
Title: Relapse-Prevention Booklets as an Adjunct to a Tobacco Quitline
Brief Title: Relapse-Prevention Booklets as an Adjunct to a Tobacco Telephone Helpline("Quitline")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-15725
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Smoking Cessation
Keywords: self help; smoking cessation; cancer prevention
MeSH Terms: conditions — Smoking Cessation | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (UC) (Active Comparator): Receive Quitline services
  Interventions: Behavioral: Smoking Cessation
- Repeated Mailings (RM) (Active Comparator): Receive the 8 Forever Free booklets sent by mail at regular intervals over a period of 12 months
  Interventions: Behavioral: Smoking Cessation
- Massed Mailings (MM) (Active Comparator): Receive all 8 booklets in a single mailing
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Behavioral: Smoking Cessation — Approximately 3400 quitline clients will be randomized to one of three conditions at the point of their 2-week follow-up call.
  Other Names: Quitline; NYSSQL; relapse-prevention; Forever Free

SUMMARY:
The study primary purpose is smoking relapse prevention. This study is a collaboration between researchers who developed the relapse-prevention intervention, at the H. Lee Moffitt Cancer Center in Tampa, Florida, and those associated with the "New York State Smokers' Quitline" (NYSSQL), at Roswell Park Cancer Institute in Buffalo, New York.

DETAILED DESCRIPTION:
In this study, approximately 3400 quitline clients will be randomized to one of three conditions at the point of their 2-week follow-up call. One-third will be randomized to a Usual Care (UC) condition, which will receive regular quitline services. One-third will be randomized to a Repeated Mailings (RM) condition, which will receive the 8 Forever Free booklets sent by mail at regular intervals over a period of 12 months. And one-third will be randomized to a Massed Mailings (MM) condition, which will receive all 8 booklets in a single mailing.

ELIGIBILITY:
Inclusion Criteria:

* referrals from the New York State Smokers' Quitline
* at least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3830 (Actual)
Dates: Start 2008-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
7-Day Point-Prevalence Abstinence at Each Follow-up Point | 24 months
  To test the effectiveness of a self-help, relapse-prevention intervention (Forever Free booklets) as an adjunct to a state telephone quitline

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States